CLINICAL TRIAL: NCT06251999
Title: Efficacy and Safety of Fospropofol Disodium Sedation for Same-day Bidirectional Endoscopy in Elderly Patients: a Prospective, Single-center, Randomized, Double-blind, Non-inferiority Trial
Brief Title: Efficacy and Safety of Fospropofol for Same-day Bidirectional Endoscopy in Elderly Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Xiaofeng WANG, Principal investigator, Shanghai 6th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XWANG
Record Dates: First submitted 2024-01-21; First posted 2024-02-09 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Elderly Patients
Keywords: fospropofol; propofol; sedation; elderly; bidirectional endoscopy
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fospropofol (Experimental)
  Interventions: Drug: fospropofol sedation
- propofol (Placebo Comparator)
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: fospropofol sedation — Fospropofol sedation for same-day bidirectional endoscopy in elderly patients
  Arms: fospropofol
Drug: Propofol — propofol
  Arms: propofol

SUMMARY:
Introduction: Fospropofol disodium is a novel prodrug that has improved pharmacokinetic and pharmacodynamic properties compared with propofol. This trial aims to compare the efficacy and safety of fospropofol versus propofol sedation for same-day bidirectional endoscopy in elderly patients.

Methods and analysis: This is a prospective, single-center, double-blind, randomized, propofol-controlled, non-inferiority trial. A total of 256 adult patients scheduled for same-day bidirectional endoscopy under sedation will be randomly allocated, in a 1:1 ratio, to a fospropofol group or a propofol group (n=128 in each group). All patients will receive analgesic pretreatment with sufentanil 5 μg. Two minutes later, an initial bolus dose of fospropofol 6.5 mg/kg or 1.5 mg/kg propofol and supplemental doses of fospropofol 1.6 mg/kg or 0.5 mg/kg propofol will be titrated as needed to the target sedation levels during the procedures. The primary outcome is the success rate of same-day bidirectional endoscopy. Secondary outcomes include the time to successful induction of sedation, duration, time to being fully alert, time to patient discharge, endoscopist satisfaction, patient satisfaction, and the top-up frequency and dosage of sedative medications. The safety endpoints consist of adverse events (AEs) concerning cough reflex, gag reflexes, body movement, muscular tremor, pain on injection. Sedation-related AEs, including episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia, will be also recorded. Data will be analyzed on the intention-to-treat basis.

Discussion: The investigators hypothesize that the efficacy and safety of fospropofol sedation for elderly patients undergoing same-visit bidirectional endoscopy will not be inferior to that of propofol. The findings will provide daily practice of sedation regimens for same-day bidirectional endoscopy in elderly patients.

ELIGIBILITY:
Inclusion Criteria:

* 65 years or older
* American Society of Anesthesiologists (ASA) physical status I to III
* Body mass index (BMI) 18-30 kg/m2
* Scheduled for same-day bidirectional endoscopy under sedation

Exclusion Criteria:

* Severe cardiovascular, pulmonary, renal, or liver diseases
* Previous hypotension (systolic blood pressure ≤90 mmHg), bradycardia (heart rate <50 beats/min), or hypoxemia (SpO2 <90%)
* Neurocognitive or psychiatric disorders
* Contraindications to gastroscopy (gastric retention, long-term aspirin administration, etc.)
* Hypersensitivity to study medications
* Drug or alcohol misuse
* Definite upper respiratory tract infection
* Refusal for participation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2024-08-01 (Estimated); Primary Completion 2027-05-31 (Estimated); Study Completion 2028-08-31 (Estimated)

PRIMARY OUTCOMES:
The success rate of same-day bidirectional endoscopy | Immediate time after sedation emergence
  The success rate of the gastrointestinal endoscopy was assessed according to the following criteria : 1) completion of the gastrointestinal endoscopy; 2) no need for rescue sedative/anesthetic, which means the top-up doses of the experimental drugs were administered no more than five times within any 15-min window from the initial administration to the end of the procedure.

SECONDARY OUTCOMES:
The time to successful induction of sedation | Immediate time after sedation emergence
  the time counted from the start of drug administration to the achievement of a sedation score (MOAA/S ) ≤ 1
Time to being fully alert | Immediate time after sedation emergence
  the time from gastrointestinal endoscopy extraction or/and the time from the last drug administration to a MOAA/S score of 5 on three consecutive measurements;
Time to patient discharge | Immediate time of hospital discharge
  Time to patient discharge
Endoscopist's satisfaction questionnaire | Immediate time after sedation procedure completion
  Endoscopist's satisfaction
Patient's satisfaction questionnaire | Immediate time of hospital discharge
  Patient's satisfaction
The top-up frequency and dosage of sedative medications | Immediate time after sedation emergence
  The top-up frequency and dosage of sedative medications
Incidence of adverse events (AEs) at timepoint 1 | baseline (Prior to sedation)
  Episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia.
Incidence of adverse events (AEs) at timepoint 2 | Intraoperative (during sedation)
  Episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia.
Incidence of adverse events (AEs) at timepoint 3 | Intraoperative (the timepoint of sedation emergence)
  Episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia.
Incidence of adverse events (AEs) at timepoint 4 | 15 min in post-anesthesia care unit
  Episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia.
Incidence of adverse events (AEs) at timepoint 5 | 30 min in post-anesthesia care unit
  Episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia.
Incidence of adverse events (AEs) at timepoint 6 | Immediate time of hospital discharge
  Episodes of desaturation, severe desaturation (SpO2 < 90%), hypotension, severe hypotension (decrease in mean blood pressure ≥30% of baseline), and bradycardia.

IPD SHARING:
Plan to Share IPD: No